CLINICAL TRIAL: NCT00524173
Title: Tenofovir Disoproxil Fumarate Alone Versus Its Combination With Emtricitabine for Treatment of Chronic Hepatitis B
Brief Title: Tenofovir Alone Versus Tenofovir With Emtricitabine to Treat Chronic Hepatitis B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070207; 07-DK-0207
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-03-16

CONDITIONS: Hepatitis B
Keywords: Emtricitabine; Tenofovir; Antiviral Therapy; Hepatitis B; HBV
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenofovir only (Active Comparator): Tenofovir 300mg by mouth daily for 192 weeks
  Interventions: Drug: Tenofovir
- Tenofovir & emtricitabine (Experimental): Tenofovir 300mg in combination with emtricitabine 200mg by mouth daily for 192 weeks
  Interventions: Drug: Tenofovir & Emtricitabine

INTERVENTIONS:
Drug: Tenofovir & Emtricitabine
  Arms: Tenofovir & emtricitabine
Drug: Tenofovir
  Arms: Tenofovir only

SUMMARY:
This study will test whether the combination of two medications, tenofovir and emtricitabine, are safer and more effective for treating chronic hepatitis B than tenofovir alone. Chronic hepatitis B is a liver disease caused by infection with the hepatitis B virus. Several medications, including standard and pegylated interferon and the anti-viral drugs lamivudine, adefovir, entecavir and telbivudine, are currently used to treat the disease. Problems are associated with all of these agents, however, including development of viral resistance with long-term therapy of the anti-virals. Since many patients require long-term therapy to prevent their disease from worsening, a major goal of new approaches to treatment is to prevent the development of viral resistance. Combination treatment has been shown to be an effective strategy in preventing this resistance.

Tenofovir is an anti-viral drug approved for use in patients with HIV infection. In small studies in patients infected with both HIV and hepatitis B, tenofovir lowered the level of hepatitis B virus in the blood, with no viral resistance reported when used for up to 5 years. Emtricitabine is an anti-viral drug similar to lamivudine and is effective at lowering viral load and improving liver damage.

Patients 18 years of age and older with chronic hepatitis B may be eligible for this study. Participants are admitted to the NIH Clinical Center for a complete medical history and examination, including blood and urine tests, chest X-ray, electrocardiogram, abdominal ultrasound, Fibroscan (ultrasound exam of the liver that measures the amount of scarring), bone mineral density scan and liver biopsy. They are then randomly assigned to take combination treatment with tenofovir plus emtricitabine or tenofovir alone for at least 48 weeks. During the treatment period, patients visit the Clinical Center for blood tests and a physical examination every 2 weeks for the first month and then every 4 to 12 weeks. After 48 weeks, patients are readmitted to the Clinical Center for a complete evaluation that includes all the tests done at the start of therapy, including a liver biopsy. Patients who seem to have improved with treatment may continue therapy for up to 192 weeks, when they are again admitted to the Clinical Center for a complete medical evaluation and liver biopsy. Patients whose condition has not improved after 48 weeks of treatment have their treatment changed or stopped and continue to have regular outpatient clinic visits for 24 more weeks.

DETAILED DESCRIPTION:
Chronic hepatitis B is a major cause of cirrhosis, end-stage liver disease and hepatocellular carcinoma and affects approximately 1.25 million Americans. Six medications have been licensed for use in chronic hepatitis B in the United States, but their relative benefit and long-term efficacy remain unclear. In previous studies, we have shown that maintained suppression of hepatitis b virus DNA (HBV DNA) can be achieved with nucleoside analogues and that suppression is associated with marked improvements in disease. In this randomized study, we propose to evaluate long-term therapy with tenofovir alone or in combination with emtricitabine (FTC). Forty treatment-naive patients with chronic hepatitis B will be enrolled in the primary study. After medical evaluation and liver biopsy, patients will be stratified by hepatitis B e antigen (HBeAg) status and randomized to receive either tenofovir alone or in combination with FTC. Treatment will be continued long-term (at least four years) and patients will be carefully monitored for side effects, serum aminotransferase and HBV DNA levels. Patients will undergo repeat liver biopsy and assessment of antiviral resistance at 1 and 4 years. The primary endpoint of therapy will be the maintained suppression of HBV DNA to below 10(2) copies/ml (lower limit of detection of current assays). The study will assess the relative efficacy and safety of combination versus mono-therapy. A separate group of 60 previously treated patients will also be enrolled and randomized to mono- or combination-therapy to assess the safety profile of these agents. The primary analysis will be conducted on the entire study cohort.

ELIGIBILITY:
* INCLUSION CRITERIA (nucleoside analogue-naive subjects):
* Age greater than 18 years and older, male or female.
* Known serum HBsAg positivity for 24 weeks.
* Detectable HBV DNA greater than 10(4) IU/ml. For patients with cirrhosis HBV DNA greater than 10(3) IU/ml
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels 1.5 times the upper limit of normal (for ALT: greater than or equal to 62 U/L and for AST greater than or equal to 46 U/L) based on at least two determinations taken at least one month apart during the 24 weeks before study entry; no ALT requirement for patients with cirrhosis.
* Liver biopsy within 2 years of entry that is consistent with chronic hepatitis and with a histology activity index (HAI) score of 4 or more (scores range from 0-18) and an Ishak fibrosis score of at least 1 (scores range from 0-6). For patients who have had a liver biopsy at another institution, slides must be obtained for reading and scoring at the NIH.
* Written informed consent.

INCLUSION CRITERIA SALVAGE STUDY (nucleoside analogue experienced subjects):

* Age >18 years and older, male or female
* Known serum HBsAg positivity for 6 months
* Detectable HBV DNA >10(2) IU/ml.
* Liver biopsy within 5 years of entry that is consistent with chronic hepatitis
* Written informed consent

INCLUSION CRITERIA: SALVAGE STUDY (relapsers)

* Age greater than 18 years and older, male or female.
* Known serum HBsAg positivity for 6 months.
* Detectable HBV DNA greater than 10(3) IU per milliliter.
* Liver biopsy within 5 years of entry that is consistent with chronic hepatitis.
* Written informed consent.

Serum ALT or AST levels 1.5 times the upper limit of norma (ULN) (for ALT: greater than 62 U/L and for AST: greater than 46 U/L) based on at least two determinations taken at least 2 weeks apart.

EXCLUSION CRITERIA:

* Previous or current treatment with tenofovir or emtricitabine.
* Co-infection with hepatitis delta virus (HDV) as defined by the presence of anti-HDV in serum and/or HDV antigen in the liver.
* Co-infection with hepatitis c virus (HCV) as defined by the presence of HCV RNA in serum.
* Co-infection with HIV as defined by the presence of anti-HIV in serum.
* Decompensated liver disease as defined by serum bilirubin greater than 2.5 milligram per deciliter (with direct bilirubin greater than 0.5 milligram per deciliter), prothrombin time of greater than 2 seconds prolonged, a serum albumin of less than 3 grams per deciliter, or a history of ascites, variceal bleeding or hepatic encephalopathy.
* Presence of other causes of liver disease (i.e. hemochromatosis, Wilson disease, alcoholic liver disease, nonalcoholic steatohepatitis, alpha-1anti-trypsin deficiency).
* A history of organ transplantation or in the absence of organ transplantation, any immunosuppressive therapy requiring the use of more than 5 milligrams of prednisone (or its equivalent) daily.
* Significant systemic illness other than liver diseases including congestive heart failure, renal failure, chronic pancreatitis, diabetes mellitus with poor control that in the opinion of the investigator may interfere with therapy.
* Pregnancy or inability to practice contraception in patients capable of bearing or fathering children and lactating women.
* Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver that is suggest of HCc, or an alpha-fetoprotein level of greater than 500ng/mL.
* History of clinically apparent pancreatitis or evidence of subclinical pancreatitis as shown by serum amylase values twice the upper limits of the normal range and abnormalities of the pancreas on CT or other imaging studies of the abdomen.
* Sensory or motor neuropathy apparent from medical history and physical examination.
* Creatinine clearance less than 50 ml/min, serum creatinine greater than 1.3 mg/dl or urine protein greater than 1 gram/24 hours; creatinine clearance will be determined on the average of two 24 hour urine specimens. Accuracy of collection will be ensured by documenting appropriate total creatinine excretion in the 24 hour urine specimen (15mg/kg) and correcting for the patient's age, gender and body surface area.
* Concurrent use of nephrotoxic agents (e.g. aminoglycosides, amphotericin B, vancomycin, foscarnet, cis-platinum, pentamidine, nonsteroidal anti-inflammatory agents) or competitors of renal tubular excretion (e.g. probenecid) within 2 months prior to study screening or the expectation that the subject will receive these during the course of the study.
* History of hypersensitivity to nucleoside analogues.
* Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, personality disorder that, in the investigator's opinion, might interfere with participation in the study.
* History of renal tubular acidosis.
* History of malignancy or treatment for a malignancy within the past 5 years.
* Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study for at least 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08-29; Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lai CL, Shouval D, Lok AS, Chang TT, Cheinquer H, Goodman Z, DeHertogh D, Wilber R, Zink RC, Cross A, Colonno R, Fernandes L; BEHoLD AI463027 Study Group. Entecavir versus lamivudine for patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1011-20. doi: 10.1056/NEJMoa051287. PMID 16525138
- [Background] Hadziyannis SJ, Tassopoulos NC, Heathcote EJ, Chang TT, Kitis G, Rizzetto M, Marcellin P, Lim SG, Goodman Z, Wulfsohn MS, Xiong S, Fry J, Brosgart CL; Adefovir Dipivoxil 438 Study Group. Adefovir dipivoxil for the treatment of hepatitis B e antigen-negative chronic hepatitis B. N Engl J Med. 2003 Feb 27;348(9):800-7. doi: 10.1056/NEJMoa021812. PMID 12606734
- [Background] Dienstag JL, Schiff ER, Wright TL, Perrillo RP, Hann HW, Goodman Z, Crowther L, Condreay LD, Woessner M, Rubin M, Brown NA. Lamivudine as initial treatment for chronic hepatitis B in the United States. N Engl J Med. 1999 Oct 21;341(17):1256-63. doi: 10.1056/NEJM199910213411702. PMID 10528035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the Protocol Section (35) conflicts with the number of participants Started in the Participant Flow module (32). Two participants failed screening and one participant declined participation after enrollment and prior to beginning treatment.
Groups:
- Tenofovir Only: Tenofovir 300mg by mouth daily for 192 weeks
  Tenofovir
- Tenofovir & Emtricitabine: Tenofovir 300mg in combination with emtricitabine 200mg by mouth daily for 192 weeks
  Tenofovir & Emtricitabine
Period: Overall Study
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
Started | 17 | 15
Completed | 12 | 13
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Had not reached endpoint at study close | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.65 (16.66) | 39.47 (12.67) | 39.56 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 15 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 10 | 20
  Black | 4 | 0 | 4
  White | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Hepatitis b Virus (HBV) DNA <1000 IU/ml at Week 48
Description: Number of subjects whose serum HBV DNA level was <1000 IU/ml at Week 48
Time Frame: At Week 48
Population: The number of participants analyzed (25) is smaller than the number of participants started (32). One participant was lost to follow-up prior to the endpoint, one died prior to the endpoint, and 5 had not reached the endpoint at study closure. Patients were transferred to another protocol to continue treatment as appropriate.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
Number analyzed (Participants) | 12 | 13
Participants | 11 | 13

2. Primary Outcome: Number of Participants With HBV DNA <1000 IU/ml at Week 192
Description: Number of participants whose serum HBV DNA level was <1000 IU/ml at Week 192
Time Frame: At Week 192
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
Number analyzed (Participants) | 12 | 13
Participants | 12 | 12

3. Secondary Outcome: Number of Participants With Normalized Alanine Aminotransferase (ALT)
Description: Number of participants whose serum ALT levels were measured within normal limits.
Time Frame: 192 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
Number analyzed (Participants) | 12 | 13
Participants | 8 | 13

4. Secondary Outcome: Number of Participants With Loss of HBsAg
Description: The number of participants whose serum hepatitis B surface antigen was no longer detectable.
Time Frame: 192 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
Number analyzed (Participants) | 12 | 13
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 192 weeks
Arm/Group | Tenofovir Only | Tenofovir & Emtricitabine
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/15
Other Adverse Events (participants affected / at risk) | 7/17 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir Only (N=17) | Tenofovir & Emtricitabine (N=15)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Only (N=17) | Tenofovir & Emtricitabine (N=15)
Aalanine aminotransferase >5xULN (Hepatobiliary disorders) | 2 | 3
Aspartate Aminotransferase > 5xULN (Hepatobiliary disorders) | 1 | 3
Creatine kinase > 4xULN (Musculoskeletal and connective tissue disorders) | 3 | 3
Neutrophils (<750mm^3) (Blood and lymphatic system disorders) | 1 | 0
Serum amylase >2xULN (Endocrine disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT00524173/Prot_SAP_000.pdf